ID: GCO 21-0434 Dual JAK1/TYK2 Inhibitor for Cicatricial NCT05076006 Alopecia

#### 

GCO# 21-0434 IRB# 21-00017

Form Version Date: May 8, 2023

#### **STUDY INFORMATION:**

Study Title: A Pilot Study to Assess Safety and Biomarker Responses of the Dual JAK1/TYK2 Inhibitor (Brepocitinib) for Cicatricial Alopecia

Principal Investigator (Head Researcher): Emma Guttman-Yassky, MD, PhD

Physical Address: Icahn School of Medicine at Mount Sinai

Departments of Dermatology and the Immunology Institute

5 East 98 Street, 5th Floor, Box 1048

New York, NY 10029

Mailing Address: 5 East 98 Street, 5th Floor, Box 1048

New York, NY 10029

**Phone:** 212-241-3288

#### **SUMMARY OF THIS RESEARCH STUDY:**

In medicine there are many unanswered questions. A research study is when scientists try to answer a question about something that we don't know enough about. Participation in a research study may or may not directly help you or others. Participation is entirely voluntary. It is completely up to you whether or not you take part. You can also change your mind at any time and it will not affect your ability to get medical care within the Mount Sinai Health System.

The purpose of this research study is to evaluate the effectiveness and safety of brepocitinib (PF-06700841 which is a type of medication classified as an oral JAK inhibitor) and the effects of brepocitinib in skin and blood in persons with Cicatricial Alopecia (CA). CA, also known as scarring alopecia, is a type of alopecia in which hair follicles are irreversibly destroyed. CA leads to scarred areas, most commonly on the scalp, that cannot re-grow hair.

If you choose to participate, you will be asked to read and sign this consent form before any study tests are done. This study includes a screening period, a Treatment Period, an End of Treatment Visit, and a Follow-up Visit. Each period is explained in this consent form in the order that they will be completed. This study will involve physical examinations, visual assessments, laboratory tests, photographs of your scalp, eyebrows, eyelashes, and fingernails, and skin biopsies. Some of these lab samples may be stored. If you are eligible for this study, you will receive either the study drug being tested, called brepocitinib, or placebo (pills without active ingredients for 24 weeks, and then all subjects will receive brepocitinib for another 24 weeks.

------FOR IRB USE ONLY-------ev 1.16.19



### 


#### GCO# 21-0434 IRB# 21-00017

You will participate in the study for approximately one year. There are 15 in-clinic visits. You will be compensated for participating in the study.

In previous brepocitinib studies, the negative effects that were reported in more than 5% (1 in 20) of study participants were upper respiratory tract infection, common cold (including inflammation of the tissue lining the sinuses, nasal passages and back of the throat), bronchitis (inflammation of the bronchial tubes that could lead to shortness of breath), headache, nausea, diarrhea, acne and decreased white blood cells, although the association with study drug is unclear.

Participating in this research may not benefit you directly. The findings from this study may help to identify new therapies for this disease. You may also benefit from participation in this research if the study drug improves your condition, or improves your quality of life.

Instead of participating in this research, you may decide to pursue other clinical trials or choose no treatment. There currently are no approved treatments for Cicatricial Alopecia.

If you are interested in learning more about this study, please continue to read below.

#### PARTICIPATION IN THIS RESEARCH STUDY:

This research study will be fully explained to you by a member of the study team. Feel free to ask all the questions you want before you make a decision about whether or not to participate. Any new information that develops during this research study that might make you change your mind about participating will be given to you promptly.

You may qualify to take part in this research study because you have Cicatricial Alopecia and are at least 18 years old.

Funds for conducting this research are provided by Pfizer Inc. The study doctor/institution are being paid by Pfizer Inc. for the work done for this study.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### LENGTH OF TIME AND NUMBER OF PEOPLE EXPECTED TO PARTICIPATE:

Your participation in this research study is expected to last 56 weeks. There will be 15 total visits that include a screening visit, Phase I (visits 2-7), Phase II (visits 9-14), and a four week follow-up visit. The

ev 1.16.19

Effective Date: 5/30/2023 End Date:3/27/2024 -----FOR IRB USE ONLY-----

### ****


#### GCO# 21-0434 IRB# 21-00017

number of people expected to take part in this research study at Icahn School of Medicine at Mount Sinai is approximately 50.

#### **DESCRIPTION OF WHAT'S INVOLVED:**

If you agree to participate in this research study, the following information describes what may be involved.

In addition to the visits listed, the study doctor may ask you to come in for extra visits if necessary to protect your well-being. A description of each test, procedure, or assessment is provided in this consent.

# Screening Visit (should take between 1-2 hours):

- Demographic questions
- Medical history
- Physical exam
- Electrocardiogram (also called an ECG or EKG) This test measures the electrical activity of your heart. Sticky pads connected by wires to the ECG machine will be placed on your skin.
- Vital signs (blood pressure, heart rate)
- Height and weight
- Blood draw (about 6 teaspoons) and urine collection (about 3 teaspoons) including:
  - Safety tests
  - Tests for hepatitis B, hepatitis C, human immunodeficiency virus (HIV), and tuberculosis (TB)
  - o Pregnancy test: this will be tested only if you are a female who can physically become pregnant
- Examination of your scalp, eyebrows, eyelashes and fingernails
- You will discuss with a member of the study team and agree on the type of birth control that you will use throughout the study and for 28 days after your last dose of tablets (only for women who are physically able to have children)

If you continue to qualify for the study, you will return for a Baseline visit. You will be given your study drug along with dosing instructions. All subjects will take their assigned study drug once daily as 5 tablets (one 25 mg tablet and four 5 mg tablets) for a total of 45 mg daily.

The study group to which you are assigned will be chosen by chance, like pulling names out of a hat. Neither you nor the study doctor will choose whether you receive brepocitinib or placebo (inactive substance that looks like the brepocitinib). You will have a three in four chance of being given brepocitinib. Neither you nor the study doctor will know which you are getting; however, this

-----FOR IRB USE ONLY------



# 


#### GCO# 21-0434 IRB# 21-00017

information could be obtained in an emergency. Study drug will not be made available to you after the study ends. At Week 24, if you were initially receiving placebo, you will begin treatment with brepocitinib, or if you were initially receiving brepocitinib, you will continue to receive brepocitinib.

You will be asked to return to the study site for additional visits every 4 weeks through Week 52. Your Baseline visit will last approximately 1 ½ hours, Weeks 24 and 48 will take approximately 2 ¼ hours, and other visits will take about 45 minutes each.

The following procedures will be done at <u>each</u> visit:

- We will ask you about any updates to your medical history and medications you are taking
- A study doctor will examine your scalp, eyebrows, eyelashes and fingernails
- Your blood pressure and heart rate will be measured.
- Blood draw (about 11 tablespoons at the Baseline visit and 3 tablespoons at each other visit) and urine collection (about 3 teaspoons) including:
  - Safety tests (you will need to fast for 8 hours before your Baseline, Week 24 and Week 48 visits)
- If you are a female of child bearing potential, a urine sample will be collected for a pregnancy test. This test must be negative to continue to qualify for this study.

The following procedures will only be performed at <u>some visits</u> as noted:

- You will be asked to fill out a short questionnaire about your overall health and quality of life (Baseline, Weeks 8, 16, 24, 32, 40, 48 and 52).
- You will be asked questions regarding past and current thoughts of suicide via the Columbia Suicide Severity Rating Scale (C-SSRS) (Baseline, Weeks 8, 16, 24, 32, 40, 48 and 52).
- You will have a blood sample drawn for:
  - o specialized tests that look at biomarkers in your blood to see how the study drug works in your body, how your body responds to the study drug, and if certain biomarkers can predict how severe the disease may be (Baseline, Weeks 12, 24, 36 and 48).
  - Pharmacokinetic (PK) tests, which evaluates how your body uses the study drug and how fast or slow the study drug moves through your body. A blood sample will be taken before you take your daily dose of tablets in the office at the Baseline, Week 24 and 48 visits. At Weeks 24 and 48 another blood sample will be collected at 30 minutes, 1 hour and 2 hours after taking your dose).
- Electrocardiogram (also called an ECG or EKG). This test measures the electrical activity of your heart. Sticky pads connected by wires to the ECG machine will be placed on your skin (Weeks 8, 16, 24, 32, 40 and 48).
  - You will undergo four punch biopsies (4.5 mm in size each) of your scalp during the study. A biopsy is a tissue sample, in this case a small skin sample, from which a lot of information can be obtained. 4.5 mm is the equivalent of the eraser on a pencil head. Each will require 2-3 stitches

------FOR IRB USE ONLY-------ev 1.16.19



### ****

GCO# 21-0434 IRB# 21-00017

that will be removed by the study doctor or study nurse 10-14 days later. At the Baseline visit, you will have 2 biopsies: one of these will be from your affected scalp skin, and the other from non-affected scalp skin. You will have an additional punch biopsy of your affected scalp skin taken at Week 24 and one at Week 48. Before the biopsy is performed, the skin will be cleaned, then disinfected and locally anaesthetized (to numb the skin). Then a cookie-cutter-like instrument is pressed into your skin to remove a small piece of tissue. You will be instructed on how to take care of the biopsy site.


• Photographs of your scalp, eyebrows/eyelashes and fingernails may be taken. The photo of your eyebrows/eyelashes will be close-up so that it will be difficult for anyone to identify you from the photos. These photographs may be used for publication in the future. All efforts will be made to photograph areas that do not include the face or any other identifying markers (tattoos). If there are any views that show your entire face or any identifying markers, they will be blacked out in any publication. You cannot participate in the trial if you do not consent for photographs to be taken. These may be taken at Baseline and every 8 weeks thereafter and at Week 52.

The treatment period will conclude at week 48, and subjects will be asked to return for a follow up visit at week 52 (end of trial) for continued observation of scalp and hair changes. At that visit we will ask you about any updates to your medical history and medications you are taking, you will be asked to complete a questionnaire about your overall health and quality of life, your scalp eyebrows, eyelashes and fingernails will be visually examined, photographs may be taken, and a blood sample will be collected for safety testing. Females of child bearing potential will be asked for a urine sample so that a pregnancy test can be performed.

If you are discontinued or decide to discontinue your participation in this study, you will be asked to have most of the procedures and assessments stated above.

To take part in this research project we will have to test your blood for evidence of HIV infection. HIV is the virus that causes AIDS. It can be transmitted through unprotected sex (vaginal, anal, or oral sex) with someone who has HIV, and through contact with blood, as in sharing needles (piercing, tattooing, drug equipment including needles used to inject drugs). HIV-infected pregnant women can transmit to their infants during pregnancy or delivery or while breast feeding. There are treatments for HIV/AIDS that can help an individual stay healthy. Individuals with HIV/AIDS can adopt safe practices to protect uninfected and infected people in their lives from becoming infected or being infected themselves with different strains of HIV.

By law, positive test results are reported to the NYS Department of Health for epidemiological (the study of the factors determining or influencing the presence or absence of disease) and Partner Notification purposes. If you wish to be tested anonymously you will be referred to a public testing center, but you

ev 1.16.19

### ****


#### GCO# 21-0434 IRB# 21-00017

will not be able to be in this study. Please know that New York State law protects the confidentiality of HIV test results and other related information. The law prohibits discrimination based on an individual's HIV status and services are available to help with such consequences. You are free to refuse this test, but if you refuse you will not be allowed to join or remain in this research project.

### For Women:

Since you are participating in a research study that involves experimental drugs or experimental treatments with potential risks to a developing fetus, it is recommended, for your protection, that you not become pregnant for the duration of the study. You should not participate if you are breastfeeding.

A blood pregnancy test will be done before you begin the study and a urine pregnancy test will be repeated at every visit

Therefore, practicing effective birth control is important. No individual birth control is 100% effective.

Recommended methods of birth control are:

- The consistent use of an approved hormonal birth control (pill/patches, rings),
- An intrauterine device (IUD),
- Contraceptive injection (Depo-Provera),
- Double barrier methods (Diaphragm with spermicidal gel or condoms with contraceptive foam),
- Sexual abstinence (no sexual intercourse) or
- Sterilization

Hormonal birth control, implants, and injections are only considered effective if used properly and started at least one month before you begin the study, continuing throughout the study and for one month after taking your last study drug dose. You should ask your study doctor if you should continue birth control for longer than 30 days after your last dose. If you are unsure whether the method of birth control you use is acceptable to use while participating in this study, you should ask your study doctor before you begin the study. If you are less than one year post-menopausal, there is the potential that you could become pregnant. If you or your partner becomes pregnant, or may be pregnant, at any time during the study, it is important that you tell your study doctor immediately. The trial drug may be stopped and a referral may be made to an obstetrician/gynecologist for follow-up. If you plan to become pregnant in the year following a clinical trial, speak with your study doctor.

Should you become pregnant, regardless of the outcome, Mount Sinai / the study team may ask for information on your pregnancy, even if you are withdrawn from the study. Your written consent will be obtained separately in the event that this happens.

IRB Approved

-----FOR IRB USE ONLY------FOR IRB USE

# 

GCO# 21-0434 IRB# 21-00017


#### For Men:

Since you are participating in a study that involves experimental drugs or experimental treatment with potential risks to a developing fetus, it is recommended that you use a condom and not impregnate a woman or donate sperm while you are taking the study drug, and for an additional 90 days after you stop taking the study drug. This is because levels of the study drug may be present in the sperm and/or seminal fluid even after you stop taking the study drug. You are encouraged to tell your female partner(s) and/or their doctor(s) that you are participating in a clinical trial.

#### **USE OF YOUR DATA AND/OR SPECIMENS:**

In the future, your identifiable information may be removed from the private information and/or samples that are collected as part of this research. After this removal, the information and/or samples could be used for future research studies or shared with other research teams for future research studies. You will not be informed of the details of specific research that is done with your medical information and biospecimens. That means that a research project might be done that you would not consent to if provided with the details of that research project.

The researchers would like to ask your permission to keep the data and specimens (like blood and tissue) collected from you during this study to use them in future research studies. Please tell us how we may use this material in future research studies.

| (1) Will y studies? | ou allow the | esearchers to store your information and/or specimens to use in future research |
|---|---|---|
| Yes | No | If no, please stop here. If yes, please continue to the next question. |
| ` / | | keep your information and/or specimens stored in a way that it is linked to he use of a code that can indicate the information came from you personally): |
| I agree to | have my info | rmation and/or specimens stored with a link to my identity |
| additiona | l information | earchers permission to <b>contact you</b> in the future to collect about you, discuss how your information and/or specimens might be used, or to pation in another research project? Please initial your choice: |
| Yes | No | |
| ` ' | _ | earchers permission to keep the information and/or specimens indefinitely and lies that are <b>directly related</b> to the purpose of the current study? |
| ev 1.16.1 | | FOR IRB USE ONLY |

# 

| GCO# 21-0434 | IRB# 21-00017 | Form Version Date: May 8, 2023 |
|---|---|---|
| Please initial you | ur choice: | |
| YesN | No | |
| use them for futu | the researchers permission to keep the information are studies that are <b>not related</b> to the purpoent area of research)? Please initial your of | - · |
| YesN | No | |
| information. This patterns etc. Do | to time researchers outside of medicine are<br>s might be in the field of anthropology, he<br>you give permission to use your informat<br>plogical sciences? Please initial your choice | uman origins, mapping human migration ion and/or specimens outside the fields of |
| YesN | No | |
| the information a (b) If the future rand/or specimens (i) If you allow explain why y Your permissis (ii) If you do not practical, the used. The I and/or speciments share identified the information Institutional Residential including people who passed. (6) Do you give presearchers, inc. | se came from, then one of the following with wed the researchers to contact you in the four identifiable information or speciment ion will be asked to use your information not give permission to be contacted in the for example, because you have moved, you institutional Review Board (IRB) will be a sens linked to your identity. The IRB can also health information without contacting on and/or specimens will not be more than the eview Board (IRB) is a committee of docuple not associated with this hospital or meanticipate in research. | lly, that will be done. is known specifically who the information ill be done: future, they may be able to contact you to is needed and what will be done with it. and/or specimens in that research project. future, or if it is found that contacting you is our identifiable data and specimens may still asked for permission to use the information give permission for researchers to use and g you, but only if it determines that sharing a a minimal risk to you or your privacy. The etors and scientists and nonscientists, edical school, whose job it is to protect tens and/or information given to other nic institutions and for profit companies, for |
| YesN | • | • |
| | FOR IRB USE ONLY | |
| ev 1.16.19 | | |

### 


GCO# 21-0434 IRB# 21-00017

| repositor | u give permission to have portions of the specimens and/or data <b>deposited in large publices</b> , (explained below) for use in research with the limits you may have chosen above? tial your choice: | c |
|---|---|---|
| Yes | No | |
| | re powerful research, it is helpful for researchers to share information they get from study mples. They do this by putting it into one or more scientific databases, where it is stored | in |

To do more powerful research, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. Researchers can then study the combined information to learn even more about health and disease. If you agree to take part in this study, some of your genetic and health information might be placed into one or more scientific databases. There are many different kinds of scientific databases; some are maintained by Icahn School of Medicine at Mount Sinai or another institution, some are maintained by the federal government, and some are maintained by private companies. For example, the National Institutes of Health (an agency of the federal government) maintains a database called "dbGaP." A researcher who wants to study the information must apply for permission to use the database. Different databases may have different ways of reviewing such requests. Researchers with an approved study may be able to see and use your

information, along with that from many other people. Researchers will always have a duty to protect your privacy and to keep your information confidential, but there are risks associated with data collection and sharing. They are described in more detail in the risks section.

#### YOUR RESPONSIBILITIES IF YOU TAKE PART IN THIS RESEARCH:

If you decide to take part in this study you will be responsible for the following things:

- While you are taking part in this study, you should not take part in another study without notifying the study doctor.
- You must follow the instructions you are given by the study doctor and study staff. If you do not follow the instructions, your visit may have to be rescheduled, or you may be discontinued from the study.
- Tell the study doctor or the study staff about all prescription and non-prescription medications, supplements, herbal preparations, or vaccines before you take them.
- Notify the study doctor or study staff if you move and provide your new address and contact information.

#### COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION:

Taking part in this research study may lead to added costs to you. Certain safety tests or assessments may uncover underlying diseases or problems that require medical attention.



------FOR IRB USE ONLY------

### 


GCO# 21-0434 IRB# 21-00017

If you agree to take part in this study, we will pay you \$175 for visit 2; \$50 for visits 3-7, 9-13, and visit 15; and \$125 for visits 8 and 14 (for a total of \$975 if you complete all study visits). You will not be compensated for the screening visit. If you do not complete this study, for any reason, you will be paid for the study visits you do complete.

Payment will be given to you in the form of a check at the end of the study (or you may request to receive this payment every 6 months). Checks require some time to be prepared and will be given to you once processed and available.

Tax law may require the Mount Sinai Finance Department to report the amount of payment you receive from Mount Sinai to the Internal Revenue Service (IRS) or other agencies, as applicable. Generally, this reporting would take place if you receive payments that equal \$600 or more from Mount Sinai in a calendar year. You would be responsible for the payment of any tax that may be due.

#### **POSSIBLE BENEFITS:**

It is important to know that you may not get any benefit from taking part in this research. Others may not benefit either. However, possible benefits may be that your CA improves or your CA flare may be shorter.

#### REASONABLY FORESEEABLE RISKS AND DISCOMFORTS:

#### Physical Risks:

In addition to these risks, this research may hurt you in ways that are not known. The unknown risks might be minor or might be major (death).

There are risks to taking part in any research study. Side effects may occur. Some of those side effects can be treated. Some side effects may go away when you stop taking the study drug. Some side effects can be mild, but others may continue longer or become permanent. Some may be life-threatening or fatal.

As this study continues, the drug manufacturer may learn more information about the study drug. You will be given new information about this study in a timely manner. This way you can decide if you want to continue to take part in this study. You may be asked to read and sign a new consent form.

## Study drug Brepocitinib Risks:

Serious or Unusual Infections

Drugs that affect the immune system such as brepocitinib may make you more likely to get infections or worsen any infection you may already have. Some infections may be serious, such as pneumonia or blood poisoning (sepsis). Most infections in clinical studies with oral brepocitinib have been mild or

------FOR IRB USE ONLY-------ev 1.16.19



### 


GCO# 21-0434 IRB# 21-00017

moderate in severity. The most common infections reported in more than 5% [1 in 20] of participants in oral brepocitinib studies were upper respiratory tract infection, nasopharyngitis (swelling of nasal passages and back of the throat), bronchitis (swelling of the bronchial tubes), sinusitis (swelling of the sinuses), headache, nausea, diarrhea, acne and decreased white blood cells. You should not start taking brepocitinib if you have any kind of infection. After starting brepocitinib, call your study doctor right away if you have any symptoms of an infection. Symptoms of an infection could include fever, weight loss, or excessive tiredness, or other symptoms specific to the site of infection, such as a persistent cough.

#### Reactivation of Viruses

Certain viruses can be stored in the body and they may reactivate (wake up) and cause negative effects, such as the chickenpox virus which causes shingles (a painful or burning skin condition), and Herpes simplex virus which causes cold sores or fever blisters in the mouth or genital ulcers. We do not know if brepocitinib could lead to the reactivation of hepatitis viruses. You will not be allowed to participate in the study if your blood tests show that you have had hepatitis types B or C viruses or if you have had history of repeated episodes of shingles (Herpes zoster virus). During the study, you should inform your study doctor (either by phone or at your next visit) if you think you may have shingles, ulcers in the genital area, or cold sores. For the same reason described above, live vaccines should not be taken prior to or after taking brepocitinib, according to the study protocol.

#### Cancer

Brepocitinib may increase the risk of certain cancers by changing the way your immune system defends against cancer. Lymphoma (blood cancer) and other cancers, including skin cancers, have occurred in patients taking medications that work in a similar way to brepocitinib. In completed brepocitinib studies, one squamous cell carcinoma of the skin and one early stage cervical cancer were reported. Most people with a history of cancer will not be eligible for this study, except for those who have had successfully treated skin cancers that were not the melanoma type and those who have had successfully treated local cancer of the cervix (the lower part of the uterus). Talk to your study doctor if you have had any type of cancer.

#### Changes in certain laboratory tests

Brepocitinib may affect your blood tests. Some changes in blood tests that have occurred in earlier studies with brepocitinib are described below. Blood tests will be checked before you start taking brepocitinib and on a regular basis throughout the study to make sure they are not changing abnormally. You will be discontinued from the study if your blood tests show abnormality which would cause concern for your continued participation in the study.

• Changes in lymphocyte counts. Lymphocytes are a type of white blood cell that help the body fight off infections and cancers. If your lymphocytes are low, you might be more likely to have an infection.

------FOR IRB USE ONLY------ev 1.16.19

Effective Date: 5/30/2023 End Date:3/27/2024

IRB Approved

# 

#### GCO# 21-0434 IRB# 21-00017

• Decreases in neutrophil counts. Neutrophils are another type of white blood cell that help the body fight off infections. If your neutrophils are low, you might be more likely to have an infection.


- Changes in platelet counts. Platelets are a type of blood cells that help blood to clot. If your platelets are low, you might be more likely to bruise or bleed. Although bleeding or bruising related to low platelets or increased clotting related to increased platelets have not been seen in previous studies with brepocitinib, there is still a potential risk that these events could happen.
- Increases in serum creatinine. Serum creatinine is a chemical that is measured in the blood to see how well your kidneys work. Increased creatinine levels in the blood may indicate that kidney function is impaired.
- Increases in serum creatine phosphokinase. Creatine phosphokinase is a protein that leaks out of muscle tissue and if the levels are high this could signify muscle injury. Very high levels of creatine phosphokinase may result in a condition called rhabdomyolysis (breakdown of muscle fibers that occurs due to muscle injury), which may lead to muscle pain, tenderness, weakness and/or kidney injury.
- Increases in hepatic transaminases. Hepatic transaminase is a chemical that is measured in the blood to see how well your liver works.
- Changes in other laboratory tests, such as your blood cholesterol or hemoglobin (red blood cells) levels may also be seen.

# Changes in Heart Rhythm (ECG- electrocardiograms)

A previous study to assess the potential for brepocitinib to affect the ECG in healthy humans showed modest changes in QT prolongation (which means the heart muscle takes longer than normal to recharge between beats). Your doctor will be monitoring your heart rhythm throughout the study with ECGs. Certain products (medicines or foods) known to affect your ECG will disqualify you from entry into the study or lead to early termination from the study if you start these products during the study. If you have questions about these products, or any new medications, talk with your study doctor. To date there have been no clinically significant reports of adverse ECG changes in humans in clinical studies with brepocitinib.

#### Risk of Allergic or Hypersensitivity Reaction

There is a chance that you may experience a local or generalized allergic reaction (also known as hypersensitivity reactions) to the study drug. One kind of allergic reaction can happen immediately (within minutes or hours) after taking study drug. This is called anaphylaxis. Symptoms of immediate allergic reaction may include skin flushing, rash or hives, sneezing, runny nose, difficulty breathing, wheezing, sudden cough, a sense of choking, sudden change in blood pressure (causing dizziness or lightheadedness), swelling around the mouth, throat, or eyes, fast pulse or sweating, abdominal cramps, diarrhea, passing out, and a sense that something bad is going to happen. The severity of this type of immediate reaction ranges from mild to severe. A mild reaction may progress to a more severe

ev 1.16.19

------FOR IRB USE ONLY------

### 


#### GCO# 21-0434 IRB# 21-00017

one, so you should contact the study personnel if you experience any new symptoms occurring within a couple of hours after study drug injection.

A severe allergic reaction requires immediate medical treatment and could result in permanent disability or death if not treated promptly. If you believe you are having a severe allergic reaction, you should immediately seek emergency medical treatment and alert the study doctor and study staff as soon as possible.

#### Bone changes

In studies with brepocitinib in juvenile rats, bone abnormalities such as malformation and/or microscopic fracture of the head of the thigh bone were noted. To date there have been no reports of bone changes associated with brepocitinib in clinical studies.

#### Other Effects

Pulmonary Embolism/Deep Vein Thrombosis -Pulmonary emboli (blood clot in the lungs) have occurred in patients taking medications that work in similar ways to brepocitinib. In ongoing brepocitinib studies, there have been events of thrombosis/pulmonary embolism, where relationship to treatment is uncertain.

If you have had a history of recent, or repeated blood clots in your legs or lungs, or have other risk factors for clotting, you may not be eligible for this study. Please let your study doctor know if you have a history of blood clots.

Events of gastrointestinal perforation (ruptured bowel) have been reported with other marketed JAK inhibitor products (the same class of drugs as brepocitinib) although the role of JAK inhibition in these events is not known. To date there have been no reports of gastrointestinal perforation in the brepocitinib clinical program.

An event of intestinal strangulation, a type of bowel obstruction where blood supply is cut off to the intestine, was observed with brepocitinib for systemic lupus. Subject recovered from event after surgery.

#### Pregnancy-related risks/Use of birth control

At this time, the effects of brepocitinib on male and female fertility, and pregnancy in humans, and effects on the fetus or a nursing child are not known. In pregnant animals, brepocitinib was associated with toxicity to the fetus which included changes in bones. In a reproduction and fertility study in male rats, no adverse effects on male fertility were noted.

In a completed brepocitinib clinical study, a cleft lip was reported in the unborn fetus of a female participant who became pregnant. The participant was also taking other medications at the same time, including an herbal supplement with a warning against use during pregnancy. Due to the investigational

------FOR IRB USE ONLY-------ev 1.16.19



#### 

#### GCO# 21-0434 IRB# 21-00017

Form Version Date: May 8, 2023 nature of brepocitinib, it should not be administered to pregnant or breastfeeding women or women of childbearing potential who are unwilling or unable to use contraception as defined in the study protocol. If you are currently pregnant, plan to become pregnant or are breastfeeding a child, you should not join this study. If you think you are pregnant, tell the study doctor immediately. Pregnancy and nonadherence to birth control will be a reason to stop taking the study drug /placebo.

If you are or become pregnant, this research may hurt your baby or your pregnancy in ways that are unknown. The unknown risks might be minor or might be major for the pregnancy. You should not become pregnant or get a woman pregnant while on this research study. Please read the acceptable methods of birth control found under the Description of What's Involved section of this document

Risk of loss of private information: this risk always exists, but there are procedures in place to minimize the risk.

Biopsy Risks: The local anesthetic injected before the skin biopsies may induce a brief burning sensation. While rare, you could have an allergic reaction to the anesthetic. Symptoms of an allergic reaction include hives or swelling of the face, lips, tongue, or throat, which may cause difficulty in breathing or swallowing. This could become life-threatening if not treated promptly. Please advise the study doctor if you have had a previous reaction to any local anesthetics.

Serious side effects from a skin biopsy are rare. The study doctor or another qualified person will use a numbing medicine (anesthetic) injection to eliminate any pain during the biopsy procedure. If you feel

pain, please tell the study doctor so he or she can inject more anesthetic to make the procedure painless. The biopsy area might feel uncomfortable after the skin sample is taken. A small scar (approximately 4.5 mm) will form once the area has healed. Occasionally, some people who do not heal well may have a thick and itchy scar that is larger than the skin biopsy site (this is called hypertrophic scar or keloid). Please let the study doctor know if you have ever developed a bad scar after a skin cut. There is also a small chance that the biopsy site may become infected which could result in pain, redness, or swelling of the area. There is also a small chance that a superficial nerve (a nerve that is responsible for the sense of touch) might be cut during the procedure. If this happens, the skin around the biopsy site may become insensitive to touch or pain. Discomfort or pain is sometimes present for a few weeks after a skin biopsy.

ECG Risks: The sticky pads placed on your skin may cause some redness or itching when the pads are removed.

Blood Draw Risks: The risks of a blood draw include pain, bruising, and the slight possibility of infection at the place where the needle goes in. Some people feel dizzy or may faint during or after a blood draw.

Group Risks: Although we will not give researchers your name, we will give them basic information such as your race, ethnic group, and sex. This information helps researchers learn whether the factors that lead to health problems are the same in different groups of people. It is possible that such findings

ev 1.16.19 IRB Approved

-----FOR IRB USE ONLY-----

### 

#### GCO# 21-0434 IRB# 21-00017

could one day help people of the same race, ethnic group, or sex as you. However, they could also be used to support harmful stereotypes or even promote discrimination.


<u>Privacy Risks</u> - Your name and other information that could directly identify you (such as address, date of birth or social security number) will never be placed into a scientific database [if true]. However, because your genetic information is unique to you, there is a small chance that someone could trace it back to you. The risk of this happening is very small, but may grow in the future. Since the database includes genetic information, a break in security may also pose a potential risk to blood relatives as well as yourself. For example, it could be used to make it harder for you (or a relative) to get or keep a job or insurance. If your private information was misused it is possible you would also experience other harms, such as stress, anxiety, stigmatization, or embarrassment from revealing information about your family relationships, ethnic heritage, or health conditions.

#### OTHER POSSIBLE OPTIONS TO CONSIDER:

You may decide not to take part in this research study without any penalty. The choice is totally up to you.

The study doctor will discuss other options and their potential risks and benefits with you before you decide whether you will take part in this study. You may also discuss your options with your regular doctor.

#### IN CASE OF INJURY DURING THIS RESEARCH STUDY:

If you are injured or made sick from taking part in this research study, medical care will be provided. Generally, this care will be billed to you or your insurance in the ordinary manner and you will be responsible for all treatment costs not covered by your insurance, including deductibles, co-payments and coinsurance. This does not prevent you from seeking payment for injury related to malpractice or negligence. Contact the investigator for more information.

#### ENDING PARTICIPATION IN THE RESEARCH STUDY:

You may stop taking part in this research study at any time without any penalty. This will not affect your ability to receive medical care at any of the Mount Sinai Health System hospitals or to receive any benefits to which you are otherwise entitled.

If you decide to stop being in the research study, contact the Principal Investigator or the research staff. For your safety, once you stop the study drug you will be asked to complete the End of Treatment Visit and Follow-Up Visit tests (as described in the description section of this form).

ev 1.16.19

-----FOR IRB USE ONLY------

### 

#### GCO# 21-0434 IRB# 21-00017

If you decide to stop being in the research study, any improvements in your CA may be lost or your CA may worsen.


If you stop being in the research study, already collected information may not be removed from the research study database and will continue to be used to complete the research analysis. You may be asked whether the study doctor can collect information from your routine medical care. If you agree, this data will be handled the same as research data.

If you decide you don't want your samples and/or data to be used for research anymore, you can contact the researcher and ask to have your samples and/or data removed from future use. Samples and data that have already been used will not be affected by your decision. Any samples and/or data that are still linked to your identity by a code the researcher has will be withdrawn so that no future sharing of your samples and/or data will take place. If your samples have already been deposited in an external repository, the study team will request that your samples be removed.

Withdrawal without your consent: The study doctor, or the institution may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the study team have not been followed, the investigator believes it is in your best interest, or for any other reason. If specimens or data have been stored as part of the research study, they too can be destroyed without your consent. More possible reasons for removal from the study include not following dosing instructions, significant laboratory test abnormalities or becoming pregnant.

#### **CONTACT INFORMATION:**

If you have any questions, concerns, or complaints at any time about this research, or you think the research has harmed you, please contact the office of the research team and/or the Principal Investigator at phone number 212-241-3288

If you experience an emergency during your participation in this research, contact 911 or go to the emergency room. Once you are able please contact the study team.

This research has been reviewed and approved by an Institutional Review Board. You may reach a representative of the Program for Protection of Human Subjects at the Icahn School of Medicine at

Mount Sinai at telephone number (212) 824-8200 during standard work hours for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You are not comfortable talking to the research team.
- You have questions about your rights as a research subject.



------FOR IRB USE ONLY------

ev 1.16.19

### 


#### GCO# 21-0434 IRB# 21-00017

• You want to get information or provide input about this research.

#### **DISCLOSURE OF FINANCIAL INTERESTS:**

Sometimes, physicians/researchers receive payments for consulting or similar work performed for industry. Effective September 2014 Mount Sinai reviews only payments to an individual totaling more than \$5,000 a year per entity when determining potential conflicts of interest. If you have questions regarding industry relationships, we encourage you to talk your physician/researcher or visit our website at http://icahn.mssm.edu/ where Mount Sinai publicly discloses the industry relationships of our faculty.

Pfizer manufactures the drug/device being tested and so has a financial interest that could be affected by the outcome of this research study.

Dr. Emma Guttman (the Principal Investigator in this study) receives financial compensation as an advisory board member for Pfizer (the study sponsor and manufacturer of the study drug). In addition, she receives financial compensation from other pharmaceutical companies that research and develop therapies used for the treatment of Alopecia. If you have questions regarding paid relationships that your physician/researcher may have with industry, we encourage you to talk with him or her, or check for industry relationships posted on individual faculty pages on our website at <a href="http://icahn.mssm.edu/">http://icahn.mssm.edu/</a>.

#### MAINTAINING CONFIDENTIALITY – HIPAA AUTHORIZATION:

As you take part in this research project it will be necessary for the research team and others to use and share some of your private protected health information. Consistent with the federal Health Insurance Portability and Accountability Act (HIPAA), we are asking your permission to receive, use and share that information.

What protected health information is collected and used in this study, and might also be shared with others?

As part of this research project, the research team at the hospital(s) involved in the research will collect your name, address, telephone/fax numbers, dates directly related to the individual (birth, admission, discharge, date of death, etc.), e-mail social security number, or photographic images

The researchers will also get information from your medical record (you will be asked to sign a release so that your primary care doctor or dermatologist can send us your medical records).

During the study the researchers will gather information by:



-----FOR IRB USE ONLY------

### 

#### GCO# 21-0434 IRB# 21-00017

 taking a medical history (includes current and past medications or therapies, illnesses, conditions or symptoms, family medical history, allergies, etc.)


- doing a physical examination that generally also includes blood pressure reading, heart rate, breathing rate and temperature
- completing the tests, procedures, questionnaires and interviews explained in the description section of this consent.
- reviewing HIV-related information, which includes any information indicating that you have had an HIV related test, or have HIV infection, HIV related illness or AIDS, or any information which could indicate that you have been potentially exposed to HIV.

# Why is your protected health information being used?

Your personal contact information is important to be able to contact you during the study. Your health information and the results of any tests and procedures done as part of this study will be used for the purpose of this study as explained earlier in this consent form. The results of this study could be published or presented at scientific meetings, lectures, or other events, but would not include any information that would let others know who you are, unless you give separate permission to do so.

The Principal Investigator may also use and share the results of these tests and procedures to treat you with others in the Mount Sinai Health System.

The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example, the School's Program for the Protection of Human Subjects is responsible for overseeing research on human subjects, and may need to see your information. If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes. If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

### Who, outside Mount Sinai, might receive your protected health information?

As part of the study, the Principal Investigator, study team and others in the Mount Sinai workforce may disclose your protected health information, including the results of the research study tests and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Principal Investigator).

IRB Approved

# 

#### GCO# 21-0434 IRB# 21-00017

- Form Version Date: May 8, 2023
- Mount Sinai laboratories who will be performing laboratory analysis for our research center.
- Our collaborator on this study, Pfizer, Inc., and their representatives or business partners, including those in other countries. Any reference to the collaborator includes their research partners and service provider including companies belonging to the collaborator, and any person or company that acquires them or the rights to the study drug (brepocitinib). The research team will send study data and results to Pfizer. Information sent to Pfizer will not include information that directly identifies you (such as your name and Social Security number) and will be coded with a participant identification number. In the future, Pfizer and their representatives, may continue to use coded health information that is collected as part of this study. Pfizer may share information from the study with regulatory agencies.
- The IRB overseeing this study: The Program for the Protection of Human Subjects
- The United States Food and Drug Administration
- The United States Department of Health and Human Services and the Office of Human Research Protection.

In all disclosures outside of Mount Sinai, you will not be identified by name, social security number, address, telephone number or any other direct personal identifier unless disclosure of the direct identifier is required by law. Some records and information disclosed may be identified with a unique code number. The Principal Investigator will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the law requires it, or rarely if the Institutional Review Board allows it after determining that there would be minimal risk to your privacy. It is possible that Pfizer or their representatives, a data coordinating office, a contract research organization, may come to inspect your

records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, when applicable, the monitors, auditors, the IRB, the Office of Human Subjects Protection (OHRP) of the Department of Health and Human Services as well as the Food and Drug Administration (FDA) will be granted direct access to your medical records for verification of the research procedures and data. OHRP and FDA are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

For how long will Mount Sinai be able to use or disclose your protected health information? Your authorization for use of your protected health information for this specific study does not expire.

#### Will you be able to access your records?

During your participation in this study, you will not be able to access your medical records. This will be done to prevent the knowledge of study results from affecting the reliability of the study. Your information will be available should an emergency arise that would require your treating physician to

ev 1.16.19

### 

#### GCO# 21-0434 IRB# 21-00017


know this information to best treat you. You will have access to your medical record and any study information that is part of that record when

the study is over or earlier, if possible. The investigator is not required to release to you research information that is not part of your medical record.

### Do you need to give us permission to obtain, use or share your health information?

NO! If you decide not to let us obtain, use or share your health information you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment or enrollment in any health plans or affect your eligibility for benefits.

# Can you change your mind?

You may withdraw your permission for the use and disclosure of any of your protected information for research, but you must do so in writing to the Principal Investigator at the address on the first page. Even if you withdraw your permission, the Principal Investigator for the research study may still use your protected information that was already collected if that information is necessary to complete the study. Your health information may still be used or shared after you withdraw your authorization if you should have an adverse event (a bad effect) from being in the study. If you withdraw your permission to use your protected health information for research that means you will also be withdrawn from the research study, but standard medical care and any other benefits to which you are entitled will not be affected. You can also tell us you want to withdraw from the research study at any time without canceling the Authorization to use your data.

If you have not already received it, you will also be given The Hospital's Notice of Privacy Practices that contains more information about how The Hospital uses and discloses your protected health information.

It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, even if your information will no longer be protected by federal regulations, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

If as part of this research project your medical records are being reviewed, or a medical history is being taken, it is possible that HIV-related information may be revealed to the researchers. If that is the case, the following information concerns you. If this research does not involve any review of medical records or questions about your medical history or conditions, then the following section may be ignored.

ev 1.16.19

# 

GCO# 21-0434 IRB# 21-00017

### • •


# **Notice Concerning HIV-Related Information**

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 306-5070. These agencies are responsible for protecting your rights.

# **ADULT PARTICIPANT:**

| • | ents your permission to take part in this<br>nealth information. A signed and dated | | |
|---|---|---|---|
| Signature of subject | Printed Name of Subject | Date | Time |

#### PERSON EXPLAINING STUDY AND OBTAINING CONSENT:

-----FOR IRB USE ONLY------

ev 1.16.19

# 

| GCO# 21-0434 | IRB# 21-00017 | Form Version | on Date: Ma | ay 8, 2023 |
|---|---|---|---|---|
| Signature of cons | sent delegate | Printed Name of consent delegate | Date | Time |
| | s required to obser | ve the consent process, it should be a<br>visually impaired, or this document a | | v |
| | accurately explaine | the information in the consent documed to, and apparently understood by, t | • | |
| Signature of Witn | ness | Printed Name of Witness | Date | Time |

------FOR IRB USE ONLY------

